CLINICAL TRIAL: NCT04823039
Title: Evaluation of Prevenar 13's Vaccine Response in Patients Hospitalized in Infectious Disease Department for Sepsis
Brief Title: Vaccine Response in Patient With Sepsis
Acronym: Vaccis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-PP-25
Record Dates: First submitted 2021-03-23; First posted 2021-03-30 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccination in patient with sepsis (Other)
  Interventions: Other: Blood sample taken

INTERVENTIONS:
Other: Blood sample taken — For patients with sepsis who require vaccination during hospitalization, we will analyze the immunogenicity of pneumococcal conjugate vaccine (PCV13) by taking blood samples

SUMMARY:
Vaccination is established as an effective means of individual and collective protection. Hospitalization is an opportunity not to be missed to catch up on vaccinations in certain fragile patients. Patients hospitalized in infectious diseases are generally treated for an acute or chronic infection that can modulate their immunity and therefore their vaccine response. Current vaccine immunogenicity data in immunocompromised patients support a lower percentage of responders than observed in immunocompetent patients.

There is little data to assess the vaccine response (VR) in patients treated for an infection (bacteremia, pneumonia, urinary tract infection, etc.). In order to respond to this problem, the investigators have chosen to evaluate the vaccine response to Prevenar 13 (PCV13), a conjugate vaccine recommended as a prime-boost since 2013, which must be followed by a vaccination at 2 months with Pneumovax, an unconjugated vaccine of 23 valences.

Anti-pneumococcal vaccine coverage in frail people (immunocompromised, heart failure, respiratory failure, kidney failure, diabetics) remains low and is estimated at less than 10% in 2011, while the bacteria is responsible for severe invasive infections.

In total, the investigators would like to study the vaccine response at 1 month of vaccination with Prevenar 13 in patients hospitalized in infectious disease for sepsis, in order to demonstrate the benefit of vaccination per hospitalization.

ELIGIBILITY:
Inclusion Criteria for all patients:

* Age ≥ 18 years old and <80 years old
* Planned length of hospital stay in infectious disease department ≥ 48 hours
* Indication for vaccination against pneumococcus according to the 2013 HAS recommendations
* Vaccination planned as part of the usual care
* Patient hospitalized for sepsis meeting the sepsis criteria according to the latest consensus of 2016 or SIRS ≥ 2 with documented infection
* Patient having signed the free and informed consent form
* Subject affiliated to social security

Inclusion Criteria for patients positive to Covid-19:

* PCR SARS-COV 2 > 0 within 28 days priodi admission and/or,
* scanner compatible with SARS-COV 2 infection.

Exclusion Criteria:

* Pregnant or breastfeeding women,
* Vulnerable people
* Pneumococcal vaccination according to the prime-boost scheme already carried out less than 5 years old
* Pneumovax vaccination <1 year
* Known hypersensitivity to the active substances or to any of the excipients or to diphtheria toxoid.
* IgG level> 1 µg / mL among more than 75% of serotypes at inclusion
* Withdrawal of consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Assess vaccine response rate at 1 month in patients with sepsis, negative to Covid-19, with an indication for pneumococcal vaccination | at 1 month
  PCV13 vaccine response rate will be measured by an ELISA method certified by WHO. Immunoglobulin G level measurements will be performed on 13 pneumococcal vaccine serotypes to analyze the vaccine response rate of patients.

SECONDARY OUTCOMES:
Evaluate cellular immunity in patients with sepsis, negative to Covid-19, with an indication for pneumococcal vaccination, at inclusion | At inclusion
  Cellular immunity will be assessed by a gamma interferon level, after non-specific stimulation of T and NK lymphocytes in the PMBC surnageant of patients cultured before vaccination (at inclusion). This level will be determined with the QFM (QuantiFERON Monitor®) test.
Identifiy the threshold of cellular immunity by the rate of gamma interferon (IFN) before vaccination (at inclusion) in patients with sepsis, negative to Covid-19, with an indication for pneumococcal vaccination | At inclusion
  Cellular immunity will be assessed by a gamma interferon level, after non-specific stimulation of T and NK lymphocytes in the PMBC surnageant of patients cultured before vaccination (at inclusion). This level will be determined with the QFM (QuantiFERON Monitor®) test.
Identify vaccine non-response risk factors at 1 month after vaccination, in patients with sepsis, negative to Covid-19, with an indication for pneumococcal vaccination | at 1 month
  Anamnestic and clinical factors of vaccine non-response will be studied
Assess the diagnostic performance (validity and reliability) of the vaccine response of PV13 at 1 month, in patients with sepsis, negative to Covid-19, with an indication for pneumococcal vaccination, assessed by an IgG VaccZymeTM anti-PCP ELISA method. | at 1 month
  Diagnostic performance (validity and reliability) of the vaccine response of PV13 will be assessed by an IgG VaccZymeTM anti-PCP ELISA method from The Binding site and the WHO validated ELISA method. Vaccinal response level from both methods will be compared.
Assess vaccine response rate at 1 month in patients with sepsis, positive to Covid-19, with an indication for pneumococcal vaccination | at 1 month
  PCV13 vaccine response rate will be measured by an ELISA method certified by WHO. Immunoglobulin G level measurements will be performed on 13 pneumococcal vaccine serotypes to analyze the vaccine response rate of patients.
Evaluate cellular immunity in patients with sepsis, positive to Covid-19, with an indication for pneumococcal vaccination, at inclusion | At inclusion
  Cellular immunity will be assessed by a gamma interferon level, after non-specific stimulation of T and NK lymphocytes in the PMBC surnageant of patients cultured before vaccination (at inclusion). This level will be determined with the QFM (QuantiFERON Monitor®) test.
Identifiy the threshold of cellular immunity by the rate of gamma interferon (IFN) before vaccination (at inclusion) in patients with sepsis, positive to Covid-19, with an indication for pneumococcal vaccination | at inclusion
  Cellular immunity will be assessed by a gamma interferon level, after non-specific stimulation of T and NK lymphocytes in the PMBC surnageant of patients cultured before vaccination (at inclusion). This level will be determined with the QFM (QuantiFERON Monitor®) test.
Identify vaccine non-response risk factors at 1 month after vaccination, in patients with sepsis, positive to Covid-19, with an indication for pneumococcal vaccination | at 1 month
  Anamnestic and clinical factors of vaccine non-response will be studied
Assess the diagnostic performance (validity and reliability) of the vaccine response of PV13 at 1 month, in patients with sepsis, positive to Covid-19, with an indication for pneumococcal vaccination, assessed by an IgG VaccZymeTM anti-PCP ELISA method. | at 1 month
  Diagnostic performance (validity and reliability) of the vaccine response of PV13 will be assessed by an IgG VaccZymeTM anti-PCP ELISA method from The Binding site and the WHO validated ELISA method. Vaccinal response level from both methods will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nice, Nice, Provence-Alpes-Côte d'Azur Region, France